CLINICAL TRIAL: NCT02750917
Title: A Comparative Study of Efficacy and Safety of Lornoxicam Versus Etoricoxib After Total Knee Arthroplasty
Brief Title: Lornoxicam Versus Etoricoxib in Postoperative Pain After Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foisor Orthopedics Clinical Hospital (Other)
Responsible Party: Principal Investigator, Munteanu Ana Maria, MD, PhD, MD, PhD, Foisor Orthopedics Clinical Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID ANALG-002-13
Record Dates: First submitted 2016-02-18; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; lornoxicam; etoricoxib; total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — lornoxicam; Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROUP LORNOXICAM (Experimental): Immediately in postoperative care unit patients received lornoxicam 8 mg PO/12 hours for 48 hours
  Interventions: Drug: Lornoxicam
- GROUP ETORICOXIB (Active Comparator): Immediately in postoperative care unit patients received etoricoxib 120 mg PO and another pill at 24 hours.
  Interventions: Drug: Etoricoxib

INTERVENTIONS:
Drug: Lornoxicam — At the end of surgery patients in group LORNOXICAM received one pill of 8 mg lornoxicam every 12 hours in the surgery day and first postoperative day.
  Other Names: XEFO RAPID; XEFO
  Arms: GROUP LORNOXICAM
Drug: Etoricoxib — At the end of surgery patients in the ETORICOXIB group received one pill of 120 mg etoricoxib at the end of surgery and a second one after 24 hours. This group also received placebo pills at 12 h, between the active pills.
  Other Names: Arcoxia; Tauxib
  Arms: GROUP ETORICOXIB

SUMMARY:
The purpose of this study is to assess efficacy and safety of lornoxicam compared with that of etoricoxib after total knee replacement.

DETAILED DESCRIPTION:
Total primary knee arthroplasty (TKA) remains a model of severe pain for major orthopedic surgery. The concept of multimodal analgesia for the postoperative pain therapy is a routine in many hospitals but the question is still under debate about the ideal combination between techniques and drugs regarding early mobilization and low risk of complications.

After obtaining Ethical Committee approval and informed consent, 110 patients American Society of Anesthesiologists score (ASA ) I-II undergoing knee replacement under spinal anesthesia were randomized to receive postoperative either lornoxicam (8 mg per os (PO) /12 hours (h) for 48 h) or etoricoxib (120mg PO/24 h for 48 h) both administered in the postoperative care unit, at the end of surgery.

The groups received postoperative analgesia when Numeric Rating Scale (NRS) over 3 with IV Perfalgan in fixed dose 1g every 8 h and morphine (loading dose 0,1mg/kg and titration until NRS under 3, followed by subcutaneous (SC) administration of ½ of the total loading dose on demand for the following 48 h).The lornoxicam group received gastric protection with IV pantoprazole.

The effectiveness was evaluated by the time from the initiation of spinal anesthesia until the first analgesic dose at NRS over 3, the total amount of morphine in the first 24 and 48 h postoperative, the side effects and necessary amount of adjuvant medication.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* weight (kilos) over 40 kg
* height (centimeters) over 155 cm
* non-anemic
* indication for primary TKA

Exclusion Criteria:

* history of asthma
* peptic ulcer
* severe hepatic or renal dysfunction
* neuropathies
* bleeding disorders
* uncooperative
* drugs abuse
* sensibility to the drugs used
* long acting nonsteroidal antiinflammatory drugs (NSAID) in the last 4 days preoperative
* cerebrovascular and peripheric vascular disease
* arterial hypertension (HTA) not adequately controlled
* congestive heart failure

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | At 48 hours postoperative
  Amount of IV and subcutaneous (SC) morphine (mg) required to reach NRS under 3

SECONDARY OUTCOMES:
Number of patients with side effects of drugs used | At 48 hours postoperative
  Number of patients with postoperative nausea and vomiting (PONV) or respiratory depression or gastric complaint or allergic reactions
Duration of analgesia | At 48 hours postoperative
  Time from spinal anesthesia until the first rescue morphine analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Ioan Cristian Stoica, Prof, Study Director — Foisor Orthopedics Clinical Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ersan O, Akkaya T, Arik E, Ates Y. Intra-articular levobupivacaine, lornoxicam and morphine analgesia after knee arthroscopy: a randomized, controlled trial. Acta Orthop Traumatol Turc. 2012;46(6):411-5. PMID 23428763
- [Background] Staunstrup H, Ovesen J, Larsen UT, Elbaek K, Larsen U, Kroner K. Efficacy and tolerability of lornoxicam versus tramadol in postoperative pain. J Clin Pharmacol. 1999 Aug;39(8):834-41. doi: 10.1177/00912709922008362. PMID 10434236
- [Background] Sener M, Yilmazer C, Yilmaz I, Caliskan E, Donmez A, Arslan G. Patient-controlled analgesia with lornoxicam vs. dipyrone for acute postoperative pain relief after septorhinoplasty: a prospective, randomized, double-blind, placebo-controlled study. Eur J Anaesthesiol. 2008 Mar;25(3):177-82. doi: 10.1017/S0265021507002827. Epub 2007 Oct 22. PMID 17953792
- [Result] Sivrikoz N, Koltka K, Guresti E, Buget M, Senturk M, Ozyalcin S. Perioperative dexketoprofen or lornoxicam administration for pain management after major orthopedic surgery: a randomized, controlled study. Agri. 2014;26(1):23-8. doi: 10.5505/agri.2014.09821. PMID 24481580
- [Result] Norholt SE, Sindet-Pedersen S, Larsen U, Bang U, Ingerslev J, Nielsen O, Hansen HJ, Ersboll AK. Pain control after dental surgery: a double-blind, randomised trial of lornoxicam versus morphine. Pain. 1996 Oct;67(2-3):335-43. doi: 10.1016/0304-3959(96)03126-0. PMID 8951927
- [Result] Buvanendran A, Kroin JS. Multimodal analgesia for controlling acute postoperative pain. Curr Opin Anaesthesiol. 2009 Oct;22(5):588-93. doi: 10.1097/ACO.0b013e328330373a. PMID 19606021